CLINICAL TRIAL: NCT05545059
Title: Effects and Safety of Sacubitril/Valsartan Versus Valsartan on Refractory Hypertension: The EOSORH Trial
Brief Title: Effects and Safety of Sacubitril/Valsartan on Refractory Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-KY-126
Record Dates: First submitted 2022-01-05; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2021-11

CONDITIONS: Resistant Hypertension
Keywords: Resistant hypertension; ambulatory blood pressure; sacubitril/valsartan; valsartan
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Amlodipine; Hydrochlorothiazide; Spironolactone; Valsartan

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sacubitril/valsartan group (Experimental): The experimental group will be sacubitril/valsartan group. Patients assigned to this group will receive sacubitril/valsartan 200mg added to existing medication regimens before randomization including amlodipine 10mg per day, hydrochlorothiazide 25 mg per day, spironolactone 20 mg per day. The initial dose of sacubitril/valsartan will be 100mg per day and will be doubled to 200mg per day after 2 weeks then maintain until the end of the 8-week treatment period.
  Interventions: Drug: Sacubitril/valsartan
- valsartan group (Active Comparator): The control group will be valsartan group, which patients will receive valsartan 160mg added to existing medication regimens before randomization including amlodipine 10mg per day, hydrochlorothiazide 25 mg per day, spironolactone 20 mg per day. The initial dose of valsartan will be 80mg per day and will be doubled to 160mg per day 2 weeks later and then maintain until the end of the 8-week treatment period.
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: Sacubitril/valsartan — In sacubitril/valsartan group, patients will receive amlodipine 10mg, hydrochlorothiazide 25 mg, spironolactone 20 mg, sacubitril/valsartan 200mg to treat. The initial dose of sacubitril/valsartan will be 100mg per day and will be doubled to 200mg per day after 2 weeks then maintain until the end of the 8-week treatment period.
  Other Names: amlodipine 10mg, hydrochlorothiazide 25 mg, spironolactone 20 mg
  Arms: sacubitril/valsartan group
Drug: valsartan — In valsartan group, patients will receive amlodipine 10mg, hydrochlorothiazide 25 mg, spironolactone 20 mg and valsartan 160mg. The initial dose of valsartan will be 80mg per day and will be doubled to 160mg per day 2 weeks later and then maintain until the end of the 8-week treatment period.
  Other Names: amlodipine 10mg, hydrochlorothiazide 25 mg, spironolactone 20 mg
  Arms: valsartan group

SUMMARY:
Resistant hypertension (RH) accounted for a considerable proportion of patients with hypertension. It has been revealed to impose certain adverse effects on the prognosis of patients with cardiovascular diseases. The antihypertensive effect of sacubitril/valsartan being fully confirmed in previous studies, there were no related randomized controlled trials (RCT) about this potency among Chinese patients with RH. The investigators designed this study to evaluated effects and safety of sacubitril/valsartan versus valsartan on Chinese patients with RH.

DETAILED DESCRIPTION:
Background Resistant hypertension (RH) accounted for a considerable proportion of patients with hypertension. It has been revealed to impose certain adverse effects on the prognosis of patients with cardiovascular diseases. The antihypertensive effect of sacubitril/valsartan being fully confirmed in previous studies, there were no related randomized controlled trials (RCT) about this potency among Chinese patients with RH.

Purpose Describing the design of the Effects of Sacubitril/valsartan Versus Valsartan on Refractory Hypertension (EOSORH) trial.

Methods and analysis This is a monocentric, randomized, parallel-group, controlled trial which will investigate the efficacy and safety of sacubitril/valsartan in the treatment of Chinese patients with RH. A total of 138 patients will be enrolled who are diagnosed with RH according to the Guidelines for Prevention and Treatment of Hypertension in China (2018 revision). After a washout period, subjects will be randomized to sacubitril/valsartan group or valsartan group in a 1:1 ratio. The primary outcome is the change in 24 hours average ambulatory systolic blood pressure (SBP) from baseline to 8 weeks after randomization, comparing the sacubitril/valsartan group with valsartan group. The secondary outcomes including change in 24 hours average ambulatory diastolic blood pressure (DBP), clinic blood pressure and series of cardiac and renal hematologic indicators. Safety endpoints will also be evaluated, covered changes in blood potassium level, renal function, hypotension, etc. Full Analysis Set (FAS), per-protocol set (PPS) and safety set (SS) will be defined. Baseline data will be analyzed by using data from FAS whereas the analysis of primary outcome will be based on FAS and PPS but the conclusions of FAS are dominant.

Ethics and dissemination The research protocol has been approved by the Ethics Committee of Sun Yat-sen Memorial Hospital, Sun Yat-sen University. This research is designed to investigate the efficacy and safety of sacubitril/valsartan in Chinese RH patients. Findings will be shared by Sun Yat-sen Memorial Hospital, policymakers and the academic community to promote the clinical pharmacal therapy of RH in China.

Discussion The effects of sacubitril/valsartan on hypertension have been widely reported by a series of large RCT in recent years, while its application in RH patients is still elusive. The study will provide a new pharmacal strategy for the treatment of RH.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of resistant hypertension
* ≥18 and ≤75 years old at the time of randomization
* Must agree to comply with all requirements and sign the informed consent form

Exclusion Criteria:

* unwilling to sign informed consent.
* Severe renal insufficiency
* Research related drug contraindications
* secondary hypertension
* Cardiovascular event
* Persistent arrhythmia, valvular heart disease, and class III-IV heart failure or left ventricular ejection fraction <45%.
* Severe liver function impairment (Child-Pugh C), biliary cirrhosis and/or cholestasis
* History of angioedema and asthma
* Woman of childbearing age who do not take effective contraceptive measures or pregnant or breastfeeding
* Allergic to drugs related to the study
* Suffering from serious tumor-related diseases, receives tumor-related treatment, or has a life expectancy of less than 2 years
* Planning to join other clinical trials
* Anticipated changes in medical conditions
* Need to take study-related drugs for reasons other than hypertension
* Suffering from other diseases that may prevent the patient from participating fully period of the study
* Other any concomitant conditions
* Must continuously take any drugs that affect the results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-09-24 (Estimated); Primary Completion 2022-10-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
the change in 24 hours average ambulatory systolic pressure from baseline to 8 weeks after randomization | 8 weeks after randomization
  the change in 24 hours average ambulatory systolic blood pressure (in mmHg) from baseline to 8 weeks after randomization

SECONDARY OUTCOMES:
Change in 24 hours average ambulatory diastolic blood pressure, daytime and night-time blood pressure and office blood pressure | 8 weeks after randomization
  Change in 24 hours average ambulatory diastolic blood pressure, daytime systolic blood pressure, night-time systolic blood pressure, daytime diastolic blood pressure, night-time diastolic blood pressure, office systolic blood pressure and office diastolic blood pressure
Change in level of cardiac marker reflecting the heart failure | 8 weeks after randomization
  serum N-terminal pro-brain natriuretic peptide (NT-proBNP in pg/ml)
Change in level of cardiac marker reflecting myocardial damage | 8 weeks after randomization
  cardiac troponin T (cTnT in pg/ml)
Change in level of novel cardiac marker reflecting the heart failure | 8 weeks after randomization
  suppression of Tumorigenicity 2 (sST2 in ng/ml)
Change in level of cardiac marker reflectting myocardial metabolism | 8 weeks after randomization
  cyclic guanosine monophosphate (cGMP in pmol/l)
Change in level of estimated glomerular filtration rate | 8 weeks after randomization
  Change in level of estimated glomerular filtration rate (eGFR in mL/min/1.73m^2).
Change in level of urinary albumin to creatinine ratio | 8 weeks after randomization
  Change in level of urinary albumin to creatinine ratio (in mg/mmol).
the control rate of blood pressure | 8 weeks after randomization
  The control rate of blood pressure. Blood pressure control was defined as a blood pressure of less than 140/90 mmHg after medical treatment.
Change in left atrium diameter determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in left atrium diameter (LA in mm) determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in left ventricular mass index determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in left ventricular mass index (LVMI in g/m^2) determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in left ventricular end diastolic volume index determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in left ventricular end diastolic volume index (LVEDVI in ml/m^2) determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in left ventricular end systolic volume index determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in left ventricular end systolic volume index (LVESVI in ml/m^2) determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in left ventricular ejection fraction determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in left ventricular ejection fraction (LVEF in %) determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in E/A determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in E/A determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.The E/A ratio is an echocardiographic index that reflects the diastolic function of the heart Under normal circumstances, E/A > 1.
Change in E/e' determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in E/e' determined by ultrasonic cardiogram and three-dimensional .The E/E' ratio is of great clinical significance in determining the diastolic function of the heart. If the E/E' ratio is <8, diastolic dysfunction can generally be ruled out. If the E/E' ratio is > 15, it generally indicates the existence of diastolic dysfunction.
Change in left ventricular overall longitudinal peak strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in left ventricular overall longitudinal peak strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in overall radial peak strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in overall radial peak strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in overall circumstantial peak strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in overall circumstantial peak strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.
Change in area strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging | 8 weeks after randomization
  Change in area strain determined by ultrasonic cardiogram and three-dimensional speckle tracking imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Dengfeng Geng, Dr., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Background] Lamirault G, Artifoni M, Daniel M, Barber-Chamoux N, Nantes University Hospital Working Group On Hypertension. Resistant Hypertension: Novel Insights. Curr Hypertens Rev. 2020;16(1):61-72. doi: 10.2174/1573402115666191011111402. PMID 31622203
- [Background] Ettehad D, Emdin CA, Kiran A, Anderson SG, Callender T, Emberson J, Chalmers J, Rodgers A, Rahimi K. Blood pressure lowering for prevention of cardiovascular disease and death: a systematic review and meta-analysis. Lancet. 2016 Mar 5;387(10022):957-967. doi: 10.1016/S0140-6736(15)01225-8. Epub 2015 Dec 24. PMID 26724178
- [Background] Kario K, Shin J, Chen CH, Buranakitjaroen P, Chia YC, Divinagracia R, Nailes J, Hoshide S, Siddique S, Sison J, Soenarta AA, Sogunuru GP, Tay JC, Teo BW, Turana Y, Zhang Y, Park S, Van Minh H, Wang JG. Expert panel consensus recommendations for ambulatory blood pressure monitoring in Asia: The HOPE Asia Network. J Clin Hypertens (Greenwich). 2019 Sep;21(9):1250-1283. doi: 10.1111/jch.13652. PMID 31532913
- [Background] Kario K, Sun N, Chiang FT, Supasyndh O, Baek SH, Inubushi-Molessa A, Zhang Y, Gotou H, Lefkowitz M, Zhang J. Efficacy and safety of LCZ696, a first-in-class angiotensin receptor neprilysin inhibitor, in Asian patients with hypertension: a randomized, double-blind, placebo-controlled study. Hypertension. 2014 Apr;63(4):698-705. doi: 10.1161/HYPERTENSIONAHA.113.02002. Epub 2014 Jan 20. PMID 24446062